CLINICAL TRIAL: NCT04502342
Title: Évaluationefficacité et tolérance d'Une médication à Base de Cosphérunate et d'un phytomédicament Antiviral Par Voie Orale en Comparaison Avec un Traitement à Base d'Hydroxychloroquine Chez Des Adultes Malades Covid-19 Sans Complications
Brief Title: Add on to Azythromycine, Phytomedicine and/or Antimalarial Drug vs Hydroxychloroquine in Uncomplicated COVID-19 Patients
Acronym: CANCOVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute for Research and Development of Medicinal and Food Plants of Guinea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDIMFPG
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: Treatment; clinical research
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Eligible consenting symptomatic patients with COVID-19 confirmed by a positive Polymerase Chain Reaction test were subjected to the 10 days of treatment allocated to each of the 3 arms of the trial. Virological clearance is assessed on days 3, 6 and 14. Side effects and the onset of COVID symptoms are evaluated throughout the trial period. Clinical, paraclinical and laboratory examinations are occasionally provided. The data are statiscally processed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine/Azythromycin (Active Comparator): Patients received Hydroxychloroquine 200 mg tablet orally 3 times daily for 10 days and Azythromycine 250 mg orally at the rate of 2 tablets the first day, then one tablet for 5 days.
  Interventions: Combination Product: Hydroxycloroquine and Azythromycine
- Cospherunate/Azithromycine (Experimental): Patients received Cospherunate (50 mg Artésunate/125 mg Amodiaquine) at the rate of 2 tablets orally twice daily for 6 days and Azythromycine 250 mg orally at the rate of 2 tablets the first day, then one tablet for 5 days.
  Interventions: Combination Product: Cospherunate/Azythromycine
- Cospherunate/Phytomedicine/Azithromycine (Experimental): Patients received Cospherunate (50 mg Artésunate/125 mg Amodiaquine) at the rate of 2 tablets orally twice daily for 6 days and Phytomedicine tablet 350 mg at the rate of 2 tablets orally twice daily for 6 days, and Azythromycine 250 mg orally at the rate of 2 tablets the first day, then one tablet for 5 days.
  Interventions: Combination Product: Cospherunate/Phytomedicine/Azythromycien

INTERVENTIONS:
Combination Product: Hydroxycloroquine and Azythromycine — dual treatment with Hydroxycloroquine and Azythromycine
  Arms: Hydroxychloroquine/Azythromycin
Combination Product: Cospherunate/Azythromycine — dual treatment with Cospherunate and Azythromycine
  Arms: Cospherunate/Azithromycine
Combination Product: Cospherunate/Phytomedicine/Azythromycien — triple treatment with Cospherunate, Asen and Azythromycine
  Other Names: Cospherunate/Asen/Azythromycine
  Arms: Cospherunate/Phytomedicine/Azithromycine

SUMMARY:
The phase II clinical trial, with three arms and at rate of 10 patients per arm, received the approval of the National Committee for Ethics and Health Research. This is a non inferiority test aimed to compare the efficacy and safety in add on to Azithromycin, an antimalarial drug, a treatment combination of the antimalrial drug with an antiviral phytomedicine versus Hydroxychloroquine in COVID-19 patients without complications.

During the treatment, viral clearance, adverse effects related to treatment, and symptoms progression will be assessed on days 3, 6 and 14. Clinical, paraclinical and laboratory tests will be performed throughout the 3-month trial. Ethical and deontological considerations will be applied.

DETAILED DESCRIPTION:
The patient who has signed the informed consent for participation in the study will be immediately taken care of by the investigating clinicians. The clinician will determine the history of the disease and identify any clinical signs shown by the patient. Clinical data will be recorded in the patient's medical file. At the end of the clinical examination, the investigating clinician will draw up the report of the biological examinations.

Laboratory examinations will be carried out according to the procedures and method by accredited laboratories in Guinea (National Institute of Public Health; Hemorrhagic Fevers Laboratory; CREMS - Kindia Laboratory; Institut Pasteur de Guinée) for the diagnosis of COVID19.

After inclusion, patients are assigned by randomization into separate treatment arms with 10 patients per arm. They remain in these treatment arms for the duration of the trial, analysis, and follow-up activities. A random sequence will be generated and implemented so as to randomize.

The treatments will be made available to investigative clinicians by the Institute for Research and Development of Medicinal and Food Plants of Guinea.

All subjects meeting the inclusion criteria will benefit from an individual file which will include data relating to general information, the complete clinical examination and the paraclinical examination. The data will be coded, entered and processed using statistical software. Data entry quality control will be performed on all files. The selected patients are distributed randomly into 3 parallel arms, each arm having a different treatment modality.

A homogeneity test on the main socio-demographic variables (age, sex, weight, hemoglobin level, etc.) will be carried out between the different treatment arms before any specific analysis. Baseline characteristics and treatment of subjects in arms 1, 2 and 3 will be presented as medians, ranges for all parameters such as clinical, anthropometric, biochemical values and as percentages or numbers for symptoms. The comparison between the three cohorts will be made using either the Anova test for continuous variables or the chi2 test for categorical variables.

The rate of change over time of virologic clearance, fever and other symptom values as well as the differences for these rates between treatment arms will be tested using mixed-effects modeling.

The duration of the trial is 20 days for each patient recruited. In anticipation of future analyzes, the biological samples will be kept at the biobank of the National Institute of Public Health of Guinea.

ELIGIBILITY:
Inclusion Criteria:

* eligible patients are symptomatic adults with COVID-19 confirmed by a positive Polymerase Chain Reaction test without complications

Exclusion Criteria:

* any patient herpersensitive to hydroxychloroquine or under antimalarial treatment in the 2 weeks preceding inclusion;
* any patient with a complication who must be taken care of in an Emergency or Intensive Care Unit;
* any patient with other acute or chronic ilnesses such as heart failure, arterial hypertension, renal failure, hepatocellular failure, tuberculosis or unable to take the oral the oral treatment;
* any patient for whom one of the treatments under study is contraindicated according to the doctor's opinion;
* pregant women;
* severe neurological manifestations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Virological clearance of throat swabs or lower respiratory tract secretions | day 3 to day 14
  Virological clearance from admission to discharge at days 3, 6 and 14

SECONDARY OUTCOMES:
Adverse effects | day 1 to day 14
  number of patients who developed treatment-related adverse effects
Worsened conditions | day 1 to day 14
  number of patients whose conditions worsened
COVID-19 symptoms | day 1 to day 14
  number of patients whose fever, cough and any other clinical sign observed on introduction have resolved

CONTACTS AND LOCATIONS:
Overall Officials: Mamadou A Baldé, Study Director — RDIMFPG
Locations (1):
- Donka; Kenien; Gbessia, Conakry, Guinea

IPD SHARING:
Plan to Share IPD: Yes
The samples stored in the biobank could be shared with other researchers with a view to in-depth analyzes in order to dig for example a posteriori on the hypotheses relating to the blood levels of the phytomedicine, hydroxychloroquine, etc., cardio-metabolic biological markers infarction, insulin sensitivity, thrombosis, specific antibodies, genetic markers, viral markers ...
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data could be available from september 30th to december 30th
Access Criteria: partnership framework established

REFERENCES:
- [Background] Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, Iosifidis C, Agha R. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). Int J Surg. 2020 Apr;76:71-76. doi: 10.1016/j.ijsu.2020.02.034. Epub 2020 Feb 26. PMID 32112977
- [Background] Mahase E. Covid-19: WHO declares pandemic because of "alarming levels" of spread, severity, and inaction. BMJ. 2020 Mar 12;368:m1036. doi: 10.1136/bmj.m1036. No abstract available. PMID 32165426
- [Background] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Background] Balde AM, Traore MS, Balde MA, Barry MS, Diallo A, Camara M, Traore S, Kouyate M, Traore S, Ouo-Ouo S, Myanthe AL, Keita N, Haba NL, Goumou K, Bah F, Camara A, Diallo MS, Sylla M, Balde ES, Diane S, Pieters L, Oulare K. Ethnomedical and ethnobotanical investigations on the response capacities of Guinean traditional health practioners in the management of outbreaks of infectious diseases: The case of the Ebola virus epidemic. J Ethnopharmacol. 2016 Apr 22;182:137-49. doi: 10.1016/j.jep.2016.02.021. Epub 2016 Feb 18. PMID 26900129
- [Background] Ayisi NK, Nyadedzor C. Comparative in vitro effects of AZT and extracts of Ocimum gratissimum, Ficus polita, Clausena anisata, Alchornea cordifolia, and Elaeophorbia drupifera against HIV-1 and HIV-2 infections. Antiviral Res. 2003 Mar;58(1):25-33. doi: 10.1016/s0166-3542(02)00166-3. PMID 12719004
- [Background] D'Alessandro S, Scaccabarozzi D, Signorini L, Perego F, Ilboudo DP, Ferrante P, Delbue S. The Use of Antimalarial Drugs against Viral Infection. Microorganisms. 2020 Jan 8;8(1):85. doi: 10.3390/microorganisms8010085. PMID 31936284
- [Background] Haladyj E, Sikora M, Felis-Giemza A, Olesinska M. Antimalarials - are they effective and safe in rheumatic diseases? Reumatologia. 2018;56(3):164-173. doi: 10.5114/reum.2018.76904. Epub 2018 Jun 30. PMID 30042604
- [Background] Das AK. Anticancer Effect of AntiMalarial Artemisinin Compounds. Ann Med Health Sci Res. 2015 Mar-Apr;5(2):93-102. doi: 10.4103/2141-9248.153609. PMID 25861527
- [Background] Gwitira I, Murwira A, Mberikunashe J, Masocha M. Spatial overlaps in the distribution of HIV/AIDS and malaria in Zimbabwe. BMC Infect Dis. 2018 Nov 27;18(1):598. doi: 10.1186/s12879-018-3513-y. PMID 30482166
- [Background] Santana Vdos S, Lavezzo LC, Mondini A, Terzian AC, Bronzoni RV, Rossit AR, Machado RL, Rahal P, Nogueira MC, Nogueira ML. Concurrent Dengue and malaria in the Amazon region. Rev Soc Bras Med Trop. 2010 Sep-Oct;43(5):508-11. doi: 10.1590/s0037-86822010000500007. PMID 21085859
- [Background] Liu DH, Liang BZ, Huang LY. [Clinical observation on the preventive effect of kangdu bufei decoction on acute severe respiratory syndrome]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2004 Aug;24(8):685-8. Chinese. PMID 15366588
- [Background] Tong X, Li A, Zhang Z, Duan J, Chen X, Hua C, Zhao D, Xu Y, Shi X, Li P, Tian X, Lin F, Cao Y, Jin L, Chang M, Wang Y. TCM treatment of infectious atypical pneumonia--a report of 16 cases. J Tradit Chin Med. 2004 Dec;24(4):266-9. PMID 15688692
- [Background] Liu BY, He LY, Liang ZW, Tong XY, Hu JQ, Jiao Q, Ni Q, Liu XM, Xie YM, Li P, Gao FZ, Wen TC, Liu WM. [Effect of glucocorticoid with traditional Chinese medicine in severe acute aespiratory syndrome (SARS)]. Zhongguo Zhong Yao Za Zhi. 2005 Dec;30(23):1874-7. Chinese. PMID 16499032
- [Background] Li Y, Liu X, Guo L, Li J, Zhong D, Zhang Y, Clarke M, Jin R. Traditional Chinese herbal medicine for treating novel coronavirus (COVID-19) pneumonia: protocol for a systematic review and meta-analysis. Syst Rev. 2020 Apr 8;9(1):75. doi: 10.1186/s13643-020-01343-4. PMID 32268923
- [Result] Efferth T, Romero MR, Wolf DG, Stamminger T, Marin JJ, Marschall M. The antiviral activities of artemisinin and artesunate. Clin Infect Dis. 2008 Sep 15;47(6):804-11. doi: 10.1086/591195. PMID 18699744
- [Result] • WHO | World Health Organization. Coronavirus (COVID-19) events as they happen [Internet]. 2020 [cited 2020 Mar 20]. Available from: https://www.who.int/emergencies/diseases/novel-coronavirus-2019/events-as-they-happen